CLINICAL TRIAL: NCT07024082
Title: Water-based Liuzijue Exercise on Childhood-onset Systemic Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assistant professor at Physical Therapy department , Faculty of Applied Medical Sciences ,Al -Zaytoonah University of Jordan, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005817
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erthematosus
Keywords: Systemic lupus erythematosus; Water-based exercise
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Land-based Liuzijue exercise (Experimental): This group includes 40 patients.Will be Performed twice a week from 9:00 to 10:00 a.m. in the rehabilitation department of Shanghai Yue-Yang Hospital under the guidance of an experienced instructor. The LG exercise program consisted of three parts: (1) Warm ups: 5-10 min of stretching and joint activity covering the limbs, neck, and trunk; (2) Land-based Liuzijue exercise: Liuzijue exercise consist of six distinct sounds (xu, he, hu, si, chui, and xi) and corresponding movements was performed with the knees in a semi-flexed position for 45 min; and the time to complete an intact Liuzijue exercise lasts 12-15 min; (3) Cool down: regulate breathing and relax muscles including flap and stretch muscles for 5-10 min.
  Interventions: Other: Land-based Liuzijue exercise
- Water-based Liuzijue exercise (Experimental): his group includes 40 patients. Water-based Liuzijue exercise will be performed twice a week, from 1:00-2:00 p.m., between June and September 2016, in the thermostatic swimming pool located at Shanghai University of Sport (Shanghai, China). The temperature of swimming pool was between 26°C and 30°C, while the temperature of air was between 30°C and 34°C, and the relative humidity was between 60% and 80%. Circulating water purification and disinfection equipment coordinated with chlorine disinfectant was used to sterilize the pool water. The participants were immersed in water to a level between their xiphisternum (lowest part of the sternum) and clavicles. Water-based Liuzijue exercise requires that participants remain awake and have eaten no sooner than 1 h prior to entering the pool to exercise. The WG exercise program consisted of three parts similar with LG:
  (1) Warm ups; (2) Water-based Liuzijue exercise; and (3) Cool down.
  Interventions: Other: Water-based Liuzijue exercise
- Control group (No Intervention): This group includes 40 patients, no exercise intervention. All participants received medical treatment.

INTERVENTIONS:
Other: Land-based Liuzijue exercise — This group includes 40 patients.Will be Performed twice a week from 9:00 to 10:00 a.m. in the rehabilitation department of Shanghai Yue-Yang Hospital under the guidance of an experienced instructor. The LG exercise program consisted of three parts: (1) Warm ups: 5-10 min of stretching and joint activity covering the limbs, neck, and trunk; (2) Land-based Liuzijue exercise: Liuzijue exercise consist of six distinct sounds (xu, he, hu, si, chui, and xi) and corresponding movements was performed with the knees in a semi-flexed position for 45 min; and the time to complete an intact Liuzijue exercise lasts 12-15 min; (3) Cool down: regulate breathing and relax muscles including flap and stretch muscles for 5-10 min.
  Arms: Land-based Liuzijue exercise
Other: Water-based Liuzijue exercise — This group includes 40 patients. Water-based Liuzijue exercise will be performed twice a week, from 1:00-2:00 p.m., between June and September 2016, in the thermostatic swimming pool located at Shanghai University of Sport (Shanghai, China). The temperature of swimming pool was between 26°C and 30°C, while the temperature of air was between 30°C and 34°C, and the relative humidity was between 60% and 80%. Circulating water purification and disinfection equipment coordinated with chlorine disinfectant was used to sterilize the pool water. The participants were immersed in water to a level between their xiphisternum (lowest part of the sternum) and clavicles. Water-based Liuzijue exercise requires that participants remain awake and have eaten no sooner than 1 h prior to entering the pool to exercise. The WG exercise program consisted of three parts similar with LG:
  (1) Warm ups; (2) Water-based Liuzijue exercise; and (3) Cool down.
  Arms: Water-based Liuzijue exercise

SUMMARY:
Systemic lupus erythematosus (SLE) is a life-long systemic autoimmune disease with a large variability in its clinical course. The onset of SLE during childhood and adolescence represents 10 to 20% of all SLE cases [1] and is associated with a more severe disease course compared to adult SLE. Due to earlier diagnosis as well as significant advances in the management of childhood-onset SLE (C-SLE), mortality rates have greatly decreased, with an estimated 5- to 10-year survival rate of over 85% [2].As a consequence, there has been a great increase in long-term co-morbidities, particularly cardiovascular disease (CVD), which is currently considered a major cause of long-term mortality in C-SLE patients [3].

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a life-long systemic autoimmune disease with a large variability in its clinical course. The onset of SLE during childhood and adolescence represents 10 to 20% of all SLE cases As a consequence, there has been a great increase in long-term co-morbidities, particularly cardiovascular disease (CVD), which is currently considered a major cause of long-term mortality in C-SLE patients. Liuzijue, which is one such traditional Chinese health exercise, is performed in expiration to produce six different sounds (xu, he, hu, si, chui, and xi) together with smooth movements of the upper and lower limbs .

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 and 15 years
* Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K score ≤ 16

Exclusion Criteria:

* Neuropsychiatry involvement, hematologic abnormalitie
* cardiovascular rhythm and conduction disorders, musculoskeletal distur- bances that precluded participation in physical exercise
* pleuritis, pericarditis, endocarditis, acute kidney failure

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2025-08-09 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory exercise test: Peak VO2 (mL/min | base line and 12 weeks
  The cardiorespiratory exercise test will be performed on a treadmill (Centurion, model 200, Micromed, Brazil), using a maximal graded exercise protocol [30]. The treadmill speed (2.0, 2.5, 3.0, 3.5, 4.0, 4.0, 4.0, 4.0, 5.0, 5.4, 5.9, 6.3, 6.3 mph), or grade (0.0, 0.0, 0.0, 0.0, 0.0, 2.5, 5.0, 7.5, 4.0, 4.0, 4.0, 4.0. 5.8%) will be increased every 1 minute. The recovery period was set at 2 minutes. Oxygen consumption (VO 2 ) and carbon dioxide output will be obtained through breath-by-breath sampling and expressed as a 30-second average using an indirect calorimetry system (Cortex, model Metalyzer III B, Leipzig, Germany).
Cardiorespiratory exercise test:Peak W (w) (working rate) (Watts) | base line and after 12 weeks
Cardiorespiratory exercise test:Chronotropic reserve (CR) % | base line and after 12 weeks
  ((CR) = (Peak HR - Resting HR/208 - (0.7 ∗ Age) - Resting HR] × 100).

SECONDARY OUTCOMES:
Functional exercise capacity | base line and after 12 weeks
  According to methods published by Ozalevli et al. [29], 30s sit-to-stand test (30 s SST) was conducted by participants. Participants sat on a 43 cm straight-backed seat, with the seat positioned against the wall to prevent falls. Participants' back was kept upright and hands were crossed so that they rested on the opposite shoulders. Before the test, participants were instructed to practice the procedure 1-2 times. During the 30 s, participants sat and stood as far as possible, and the repetitions were recorded.
Bone mineral density | base line and after 12 weeks
  BMD (g/cm 2) will be determined by dual-energy x-ray absorptiometry (DXA), using a Hologic QDR 4500 Discovery densitometer (Hologic Inc., Bedford, MA, USA). Bone area (BA) (cm 2) will be calculated using the software provided with the densitometer. Bone mass will be analyzed in the lumbar spine (lumbar vertebrae L1 to L4), total femur, and whole body.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No